CLINICAL TRIAL: NCT00912808
Title: A Study of Cholinergic Augmentation in Frequently Falling Subjects With Parkinson's
Brief Title: Cholinergic Augmentation in Frequently Falling Subjects With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Kathryn Anne Chung, Associate Professor - Neurology, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: e1784
Record Dates: First submitted 2009-06-02; First posted 2009-06-03 (Estimated); Results first posted 2011-08-15 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-04

CONDITIONS: Parkinson's Disease
Keywords: parkinsons disease; falling
MeSH Terms: conditions — Parkinson Disease | interventions — Donepezil; Sugars

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Donepezil (Experimental)
  Interventions: Drug: Donepezil
- Sugar Pill (Placebo Comparator)
  Interventions: Drug: Sugar Pill (placebo)

INTERVENTIONS:
Drug: Donepezil — donepezil, 5 mg, capsule, once a day, 3 weeks
  Other Names: aricept
  Arms: Donepezil
Drug: Sugar Pill (placebo) — sugar pill, one capsule, once a day, 3 weeks
  Arms: Sugar Pill

SUMMARY:
The purpose of this study is to find out if a medication that increases levels of a brain chemical called acetylcholine will improve balance and reduce falls in patients with parkinson's disease who have the problem of very poor balance and are frequently falling or nearly falling on a daily basis. Donepezil, a drug approved for the treatment of Alzheimer's dementia, will reduce falls in subjects with Parkinson's disease and balance impairment.

DETAILED DESCRIPTION:
This trial is a double-blinded cross-over design comparing donepezil with placebo in 40 subjects with idiopathic Parkinson's disease who report frequent falls or near falls (>2/week). The purpose of this study is to find out if a medication that increases levels of a brain chemical called acetylcholine will improve balance and reduce falls in patients with parkinson's disease who have the problem of very poor balance and are frequently falling or nearly falling on a daily basis. Donepezil, a drug approved for the treatment of Alzheimer's dementia, will reduce falls in subjects with Parkinson's disease and balance impairment.

ELIGIBILITY:
Inclusion Criteria:

* Age over 21
* Diagnosis of Parkinson's disease
* Treated with dopaminergic medication for at least 1 year

Exclusion Criteria:

* Must be ambulatory (can use walker or cane)
* No obvious remediable cause of falls
* Falls are on basis of non-CNS etiologies (cardiogenic, orthopedic, peripheral neuropathy, etc)
* Dementia present (MMSE < 25)
* Not taking cholinergic or anticholinergic medications 10 days prior to screening visit
* No Warfarin use

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2005-10; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Chung, MD, Principal Investigator — Oregon Health and Science University

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult subjects were those diagnosed with probable idiopathic PD, defined as manifesting two of three cardinal features (tremor, rigidity, bradykinesia), without any other historical or physical signs to suggest another diagnosis, and were recruited from the Oregon Health and Science University (OHSU) Movement Disorders clinic.
Pre-assignment Details: This is a cross-over treatment trial. Each drug phase, donepezil or identical placebo, lasted 6 weeks, with a three week washout period in between. In each drug phase, subjects were instructed to take one tablet (mg of donepezil or placebo) for three weeks and to increase to two tablets (10 mg) for the remaining three weeks.
Groups:
- Donepezil (6 Weeks), Washout (3 Weeks), Placebo (6 Weeks): Donepezil 5 mg qam weeks 1-3, 10 mg qam weeks 3-6 then Nothing weeks 7-9 then Placebo (sugar pill) 5 mg qam weeks 10-13, 10 mg qam weeks 14-16
- Placebo (6 Weeks), Washout (3 Weeks), Donepezil (6 Weeks): Placebo (sugar pill) 5 mg qam weeks 1-3, 10 mg qam weeks 3-6 then Nothing weeks 7-9 then Donepezil 5 mg qam weeks 10-13, 10 mg qam weeks 14-16
Period: First Intervention (6 Weeks)
Arm/Group | Donepezil (6 Weeks), Washout (3 Weeks), Placebo (6 Weeks) | Placebo (6 Weeks), Washout (3 Weeks), Donepezil (6 Weeks)
Started | 11 | 12
Received Intervention | 11 | 12
Completed | 9 | 11
Not Completed | 2 | 1
Not completed — Adverse Event | 2 | 1
Period: Washout
Arm/Group | Donepezil (6 Weeks), Washout (3 Weeks), Placebo (6 Weeks) | Placebo (6 Weeks), Washout (3 Weeks), Donepezil (6 Weeks)
Started | 9 | 11
Completed | 9 | 10
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Second Intervention (6 Weeks)
Arm/Group | Donepezil (6 Weeks), Washout (3 Weeks), Placebo (6 Weeks) | Placebo (6 Weeks), Washout (3 Weeks), Donepezil (6 Weeks)
Started | 9 | 10
Received Intervention | 9 | 10
Completed | 8 | 9
Not Completed | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: 23 participants were enrolled into the study. 3 participants screen failed.
Groups:
- Placebo (6 Weeks), Washout (3 Weeks), Placebo (6 Weeks): Placebo (sugar pill) 5 mg qam weeks 1-3, 10 mg qam weeks 3-6 then Nothing weeks 7-9 then Donepezil 5 mg qam weeks 10-13, 10 mg qam weeks 14-16
- Total: Total of all reporting groups
Arm/Group | Donepezil (6 Weeks), Washout (3 Weeks), Placebo (6 Weeks) | Placebo (6 Weeks), Washout (3 Weeks), Placebo (6 Weeks) | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 6 | 10
  >=65 years | 7 | 6 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.5 (10.2) | 66.4 (11.5) | 68.4 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 9 | 10 | 19
Region of Enrollment [Number; unit: participants]
  United States | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Fall Frequency Per Day
Description: The primary outcomes were fall frequency determined using daily event recording by the subjects onto postcards which accumulated data for six weeks per phase. Falls were defined as landing on the floor. Fall frequency is the number of reported falls divided by the number of days reported. Postcards were mailed back to the investigator weekly.
Time Frame: 6 weeks
Measure: Mean (Standard Error); unit: Number Falls/Day
Groups:
- Donepezil: Participants who received Donepezil tablet (matching 5 mg for the first 3 weeks then 10 mg for the next 3 weeks) each morning in either the first or last 6 weeks of the study.
- Placebo: Participants who received Placebo tablet (matching Donepezil) each morning in either the first or last 6 weeks of the study.
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 8 | 11
Number Falls/Day | 0.13 (0.13) | 0.25 (0.34)
Statistical Analysis 1: Comparison: Donepezil vs Placebo; Means and standard deviations were calculated to describe the subject baseline characteristics. Paired t-tests evaluated the difference between baseline and end of treatment frequency of falls. Changes post-treatment from baseline in secondary measures were also compared between the donepezil and placebo phases with paired t-tests or Wilcoxon signed rank tests when data was nonparametric. SPSS was used for the analysis; Test type: Superiority or Other; p = 0.049, t-test, 2 sided

2. Secondary Outcome: Frequency of Near Falls Per Day
Description: The secondary outcome was near fall frequency determined using daily event recording by the subjects onto postcards which accumulated data for six weeks per phase. Near falls were defined as a fall that did not land on the floor (for example grabbing a handrail or a table). Near fall frequency is the number of reported near falls divided by the number of days reported. Postcards were mailed back to the investigator weekly.
Time Frame: 6 weeks
Measure: Mean (Standard Error); unit: Number Near Falls/Day
Groups:
- Placebo: Participants who received Placebo tablet (matching Donepezil 5 mg for the first 3 weeks then 10 mg for the next 3 weeks) each morning in either the first or last 6 weeks of the study.
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 8 | 11
Number Near Falls/Day | 2.50 (4.10) | 2.04 (2.08)
Statistical Analysis 1: Comparison: Donepezil vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.27, t-test, 2 sided

ADVERSE EVENTS:
Groups:
- Donepezil Then Placebo: Donepezil 5 mg qam weeks 1-3, 10 mg qam weeks 3-6 then 3 weeks washout then Sugar pill 5 mg qam weeks 1-3, 10 mg qam weeks 3-6
- Placebo Then Donepezil: Sugar pill 5 mg qam weeks 1-3, 10 mg qam weeks 3-6 then 3 weeks washout then Donepezil 5 mg qam weeks 1-3, 10 mg qam weeks 3-6
Arm/Group | Donepezil Then Placebo | Placebo Then Donepezil
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 0/11 | 0/12

LIMITATIONS AND CAVEATS:
Small number of subjects and lack of objective measurement to quantify falls. The most difficult condition to exclude was co-existing freezing of gait.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes